CLINICAL TRIAL: NCT06144060
Title: A Multi-center, Randomized, Double-blind, Active Controlled, Parallel Groups, Phase II Study to Evaluate the Efficacy and Safety of Intravenous HRS-8427 in the Treatment of Adults With Complicate Urinary Tract Infection, Including Acute Pyelonephritis
Brief Title: A Trial of Intravenous HRS-8427 in the Treatment of Adults With Complicate Urinary Tract Infection, Including Acute Pyelonephritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-8427-202
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Patients With Complicated Urinary Tract Infection(cUTI), Including Acute Pyelonephritis(AP)
MeSH Terms: interventions — Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A：HRS-8427 (Experimental)
  Interventions: Drug: HRS -8427
- Treatment group B：HRS-8427 (Experimental)
  Interventions: Drug: HRS -8427
- Imipenem and Cilastatin Sodium (Active Comparator)
  Interventions: Drug: Imipenem and Cilastatin Sodium

INTERVENTIONS:
Drug: HRS -8427 — The dose and frequency of administration were adjusted according to the eGFR.
  Arms: Treatment group A：HRS-8427; Treatment group B：HRS-8427
Drug: Imipenem and Cilastatin Sodium — The dose and frequency of administration were adjusted according to the eGFR .
  Arms: Imipenem and Cilastatin Sodium

SUMMARY:
The Purpose of this study is to evaluate the efficacy and safety of intravenous HRS -8427 in patients with complicated urinary tract infection, including acute pyelonephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent before the study, fully understand the study and be able to complete the study according to the protocol;
2. Male and female, 18 to 75 years of age, inclusive;
3. Judged by the investigator, clinical diagnosis with cUTI or AP, expectation that the patients will require hospitalization and initial treatment with intravenous antibiotics;
4. Urine specimen with evidence of pyuria；
5. Have urine culture specimen obtained within 48 hours prior to randomization;
6. Women of childbearing potential must have a negative serum pregnancy test before first dose, must be non-lactating. Fertile female subjects or male subjects whose partner is a fertile female agree to use highly effective form of contraception, with no plan of birth, sperm/ovum donation from the time of signed ICF till 14 days after end of treatment.

Exclusion Criteria:

1. History of significant hypersensitivity or allergic reaction to any β-lactam, or any β-lactamase inhibitors;
2. Known history of immune deficiency disease or receive immunocompromising treatment;
3. Severe cardiovascular and cerebrovascular diseases with clinical significance and unstable condition or uncontrolled;
4. Known or suspected central nervous system disorder or other factors that may predispose to seizures or lower the seizures onset threshold;
5. Presence of any known or suspected disease or condition that, in the opinion of the Investigator, may confound the assessment of efficacy;
6. Uncomplicated lower urinary tract infection;
7. Suspected or confirmed urinary tract symptoms caused by acute/chronic prostatitis, orchitis, epididymitis or sexually transmitted diseases as determined by medical history and/or physical examination;
8. Patients diagnosed malignant tumors prior to randomization and currently with;
9. Systemic antimicrobial therapy other than the investigational drug need to be used during the study period, with the exception of topical or single oral dose of antifungal treatment
10. Urinary tract surgery prior to the randomization or urinary tract surgery planned during the study period;
11. Receipt of potentially effective systemic antibacterial therapy for a continuous duration of >24 hours during the previous 72 hours prior to the randomization;
12. History of pelvis or urinary tract trauma prior to the randomization;
13. Patients had severe trauma or received major surgery prior to the randomization, or surgery planned during the study period;
14. Impairment of renal function with estimated glomerular filtration rate <15 mL/min (calculated by the Modification of Diet in Renal Disease study equation);
15. Laboratory abnormalities in baseline specimens obtained at screening;
16. A QTcF interval prolongation at screening or abnormalities with clinical significance and may cause obvious safety risk to the subjects;
17. Known urine culture with at least one Gram-Negative uropathogen at ≥105 colony-forming units(CFU)/mL unsusceptible to Imipenem and Cilastatin Sodium, or only identify Gram-positive uropathogen, or confirmed fungal urinary tract infection with ≥103CFU/mL;
18. Indwelling catheter or urinary tract instrument, in the opinion of the Investigator, incapable of removal during the study period;
19. Likely to require the use of antibiotic for cUTI or AP prophylaxis after treatment;
20. Suspected of sepsis, producing life-threatening organ dysfunction;
21. Estimated survival within 6 weeks or rapidly progressive or end stage disease with high mortality rate;
22. Drug abuse prior to the randomization;
23. Participated in, any other clinical study involving the administration of active investigational or experimental medication prior to the randomization, or 5 half-lives, whichever is longer, prior to Screening;
24. In the judgment of the Investigator, other reasons unsuitable for study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Composite Response of Microbiological Eradication and Clinical Response at Test of Cure (TOC) | Test of cure (TOC; 7 days after end of treatment [EOT], equivalent to Study Day 14 to 21)

SECONDARY OUTCOMES:
Percentage of Participants With Composite Response of Microbiological Eradication and Clinical Response at Early Assessment（EA）、End of Treatment（EOT）and Late Follow-Up (LFU) | EA : Day 4、EOT: Day 7 to Day 14、LFU：Day 21 to Day 28
Percentage of Participants With Microbiological Eradication at EA（Day 4） 、EOT（End of treatment）、TOC（7 days after end of treatment） and LFU（14 days after end of treatment） | EA（Day 4） 、EOT（End of treatment）、TOC（7 days after end of treatment） and LFU（14 days after end of treatment）
Percentage of Participants With Microbiological Eradication at EA （Day 4）、EOT（End of treatment）、TOC（7 days after end of treatment） and LFU（14 days after end of treatment） Per Uropathogen | EA （Day 4）、EOT（End of treatment）、TOC（7 days after end of treatment） and LFU（14 days after end of treatment） Per Uropathogen
Percentage of Participants With Clinical Response at EA（Day 4） 、EOT（End of treatment）、TOC（7 days after end of treatment） and LFU（14 days after end of treatment） | EA（Day 4） 、EOT（End of treatment）、TOC（7 days after end of treatment） and LFU（14 days after end of treatment）
Percentage of Participants With Clinical Response at EA（Day 4） 、EOT（End of treatment）、TOC（7 days after end of treatment） and LFU （14 days after end of treatment）Per Uropathogen | EA（Day 4） 、EOT（End of treatment）、TOC（7 days after end of treatment） and LFU （14 days after end of treatment）Per Uropathogen

IPD SHARING:
Plan to Share IPD: Undecided